CLINICAL TRIAL: NCT02745327
Title: A Longitudinal Study of Childhood Intestinal Bacterial Overgrowth, Vaccine Underperformance, and Malnutrition
Brief Title: Nutrition, Overgrowth, and Vaccine Efficacy in Low-income Settings
Acronym: NOVEL
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Virginia Commonwealth University (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, William Petri, MD, Division Chief, Infectious Disease, University of Virginia
Other Study IDs: PR14083
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Small Intestine Bacterial Overgrowth
Keywords: oral vaccination; nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, stool, and urine.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the impact of small intestine bacterial overgrowth (SIBO) on childhood nutritional status, growth, and oral vaccine efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Child previously enrolled in the FIELD STUDIES protocol (enrollments in both studies may occur simultaneously)
* Mother willing to sign informed consent form.
* Healthy infant aged less than 7 days old

Exclusion Criteria:

* Parents are not willing to have child's blood drawn, oral fluid collected, urine collected, or breath testing performed.
* History of seizures, other apparent neurologic disorders, or other congenital abnormalities involving major organ systems.

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Bangladeshi infants from the low-income neighborhood of Mirpur, Dhaka
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2014-11; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Glucose-Hydrogen Breath Test | Birth to 2 years
  Test for Small Intestine Bacterial Overgrowth

SECONDARY OUTCOMES:
Fecal Regenerating Islet-Derived 1 Beta (Reg 1B) | Birth to 2 years
Fecal Myeloperoxidase | Birth to 2 years
Serum 25-OH vitamin D | Birth to 2 years
Serum Zinc | Birth to 2 years
Serum Retinol Binding Protein | Birth to 2 years
Serum Cobalamin | Birth to 2 years
Serum Albumin | Birth to 2 years
Lactulose mannitol ratio | 12 weeks of age
Serum Tetanus antibody titers | Birth to 2 years
Serum Polio antibody titers to sabin strains | Birth to 2 years
Oral fluid Tetanus antibody titers | Birth to 2 years
Height | Birth to 2 years
Weight | Birth to 2 years
Head circumference | Birth to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: William A Petri, M.D., PhD, Principal Investigator — University of Virginia
Locations (1):
- The International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Donowitz JR, Pu Z, Lin Y, Alam M, Ferdous T, Shama T, Taniuchi M, Islam MO, Kabir M, Nayak U, Faruque ASG, Haque R, Ma JZ, Petri WA Jr. Small Intestine Bacterial Overgrowth in Bangladeshi Infants Is Associated With Growth Stunting in a Longitudinal Cohort. Am J Gastroenterol. 2022 Jan 1;117(1):167-175. doi: 10.14309/ajg.0000000000001535. PMID 34693912